CLINICAL TRIAL: NCT00140036
Title: Pharmacogenomics Blood Sampling Protocol For Irinotecan/Fluorouracil/Leucovorin(CPT-11/FU/LV).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPTAIV-0020-366; A5961020
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: Blood draw

SUMMARY:
This protocol describes procedures for the collection of blood samples for the intent of determining genetic contribution to the safety and efficacy of CPT/FU/LV.

ELIGIBILITY:
Inclusion Criteria:

* Participation in studies employing treatment with irinotecan and a signed informed consent.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137
Dates: Start 2002-09; Study Completion 2005-08

PRIMARY OUTCOMES:
Correlation of genotype with safety and efficacy measures.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- United States (29):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Stamford, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Tamarac, Florida
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Annapolis, Maryland
  - Pfizer Investigational Site, Pittsfield, Massachusetts
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Hooksett, New Hampshire
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Rockville Centre, New York
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Hendersonville, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Zanesville, Ohio
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Temple, Texas
  - Pfizer Investigational Site, Newport News, Virginia
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Canada (5):
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Fleurimont, Quebec